CLINICAL TRIAL: NCT00090272
Title: A Prospective, Multicenter, Double-Blind, Randomized, Comparative Study to Evaluate the Safety, Tolerability, and Efficacy of a Single Dose of Ertapenem Sodium (MK0826) Versus Cefotetan for the Prophylaxis of Surgical Site Infection Following Elective Colorectal Surgery
Brief Title: A Single Dose of a Marketed Drug Being Studied for a New Indication to Treat Surgical Site Infection Following Colorectal Surgery as Compared to a Marketed Drug Approved for This Indication (0826-039)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0826-039; 2004_010
Record Dates: First submitted 2004-08-25; First posted 2004-08-27 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2017-02

CONDITIONS: Colorectal Surgery
MeSH Terms: interventions — Ertapenem

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: MK0826, ertapenem sodium
Drug: Comparator: cefotetan

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of a one time dose of an intravenous marketed drug being evaluated for a new indication as compared to a marketed drug already approved for the prevention of surgical site infection following colorectal surgery.

DETAILED DESCRIPTION:
The duration of treatment is 1 day.

ELIGIBILITY:
Inclusion Criteria:

Male or female patients 18 years of age scheduled to undergo elective colon or colorectal surgery by laparotomy must meet the following criteria:

* Surgery must be scheduled in advance.
* There must be adequate time to complete preoperative bowel preparation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 952 (Actual)
Dates: Start 2002-04; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Surgical site infection following elective colorectal surgery based on surgical site assessment.

SECONDARY OUTCOMES:
Microbiology of surgical site infection in pts who fail prevention or have distant site infection; Safety profile based on AE monitoring and lab results.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Itani KM, Wilson SE, Awad SS, Jensen EH, Finn TS, Abramson MA. Ertapenem versus cefotetan prophylaxis in elective colorectal surgery. N Engl J Med. 2006 Dec 21;355(25):2640-51. doi: 10.1056/NEJMoa054408. PMID 17182989
- [Background] Goldstein EJ, Citron DM, Merriam CV, Abramson MA. Infection after elective colorectal surgery: bacteriological analysis of failures in a randomized trial of cefotetan vs. ertapenem prophylaxis. Surg Infect (Larchmt). 2009 Apr;10(2):111-8. doi: 10.1089/sur.2007.096. PMID 19226203
- [Background] Itani KM, Wilson SE, Awad SS, Jensen EH, Finn TS, Abramson MA. Polyethylene glycol versus sodium phosphate mechanical bowel preparation in elective colorectal surgery. Am J Surg. 2007 Feb;193(2):190-4. doi: 10.1016/j.amjsurg.2006.08.024. PMID 17236845
- [Background] Itani KM, Jensen EH, Finn TS, Tomassini JE, Abramson MA. Effect of body mass index and ertapenem versus cefotetan prophylaxis on surgical site infection in elective colorectal surgery. Surg Infect (Larchmt). 2008 Apr;9(2):131-7. doi: 10.1089/sur.2007.034. PMID 18426345
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html